CLINICAL TRIAL: NCT05165316
Title: European Long-acting Antipsychotics in Schizophrenia Trial-II
Acronym: EULAST-II
Status: Enrolling by invitation | Type: Observational
Sponsor: Rene Kahn (Other)
Responsible Party: Sponsor-Investigator, Rene Kahn, Head of Psychiatry Department, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: 00-000
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Schizophrenia is a chronic psychiatric illness with a heterogeneous disease course, varying from periods of symptomatic remission to relapse. Relative to the wealth of scientific data on the course of schizophrenia during the two years following the first psychotic episode, the outcome of schizophrenia patients over the first decade of their illness has been studied to a lesser degree. In this follow-up cohort study the aim is to investigate the long-term outcome of schizophrenia patients who participated in the previously conducted EULAST-I clinical trial, in the first decade after being diagnosed.

DETAILED DESCRIPTION:
At this point, given the heterogeneity of published studies, it remains unclear if depot medication can reduce relapse rates and improve clinical outcome when offered to all patients in need of continuation treatment with antipsychotics. Before anyone can conclude whether or not all schizophrenia patients could benefit from a switch to depot formulations, several questions remain to be answered. Is depot medication associated with better continuation rates and outcome? How are depot medications tolerated as compared to oral medication? In order to clarify these important issues this study aims to perform a large multi-center trial in which schizophrenia patients in need of continuous treatment who are randomized 1:1:1:1 to two different depot preparations or to two different oral medications; patients will be followed up for a total of 19 months.

The primary objective of this trial is to compare all cause discontinuation rates in patients with schizophrenia randomized to oral antipsychotic medications (i.e., aripiprazole or paliperidone) versus depot antipsychotic medications (i.e., paliperidone palmitate or aripiprazole depot) over an 18 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written informed consent / have a legal representative to provide written informed consent. *
2. Having been randomized to one of the four treatment arms (aripiprazole oral, aripiprazole depot, paliperidone oral, paliperidone depot) in the 2014-002765-30 EULAST-I clinical trial or having participated in the EULAST-I naturalistic cohort study.

   * Unless prohibited by local law (e.g. due to incarceration).

Exclusion Criteria: No exclusion criteria are applicable in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with schizophrenia who participated in the previously conducted EULAST-I clinical trial. All patients who were randomized (to either aripiprazole oral, aripiprazole depot, paliperidone oral, paliperidone depot) or who participated in the naturalistic follow-up part of the EULAST-I clinical trial will be invited to participate in the current long-term follow-up cohort study (EULAST-II); this includes patients who dropped-out after randomization, patients who met All Cause Discontinuation (ACD) criteria and patients who completed the previous EULAST-I clinical trial. Patients will be over 18 years of age. The current long-term follow-up visit will take place at least three years after each patient's last visit as conducted within the EULAST-I clinical trial or the naturalistic follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To assess which baseline EULAST-I clinical trial baseline characteristics predict healthcare utilization (defined as number of days hospitalized) over a period of 3 - 10 years (since the EULAST-I clinical trial baseline visit). | 3 - 10 years (since the EULAST-I clinical trial baseline visit).

SECONDARY OUTCOMES:
To provide insight into long-term social functioning as measured through the Personal and Social Performance (PSP) scale. | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight into long-term sociodemographic outcome (living circumstances, education, marital status). | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in changes in neuropsychiatric diagnoses as measured through the Mini-International Neuropsychiatric Interview 7.0.2 (M.I.N.I. 7.0.2) since the EULAST-I clinical trial screening visit. | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in long-term outcome in quality of life as measured through the Euroqol quality of life scale (EQ-5D-5L). | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in long-term outcome in alcohol and drug use as well as smoking as measured through the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in long-term outcome of tardive dyskinesia as measured through the Abnormal and Involuntary Movement Scale (AIMS). | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in long-term outcome of extrapyramidal symptoms as measured through the St. Hans rating scale. | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight in the use of antipsychotic medication and other medication since the previous EULAST-I clinical trial. | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight into the reasons for hospitalizations since the baseline visit of the previous EULAST-I clinical trial. | 3 - 10 years (since the EULAST-I clinical trial baseline visit).
To provide insight into the incidence of suicide attempts since the baseline visit of the previous EULAST-I clinical trial | 3 - 10 years (since the EULAST-I clinical trial baseline visit).

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Hashomer The Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No